CLINICAL TRIAL: NCT04602637
Title: Training Load Management in Three Professional Tennis Players During COVID-19 Lockdown: a Case Series Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kine Kinesiologia Deportiva y Funcional (Network)
Responsible Party: Sponsor
Other Study IDs: TLT01
Record Dates: First submitted 2020-10-22; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Monitor Training Load
Keywords: training load; tennis; covid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- P1
  Interventions: Other: Training load
- P2
  Interventions: Other: Training load
- P3
  Interventions: Other: Training load

INTERVENTIONS:
Other: Training load — Monitoring training load during covid

SUMMARY:
Research describing training load management during COVID-19 enforced home training in professional tennis players is lacking. Therefore, the main objective of this case series is to describe in detail the training load management and progression of three professional tennis players before, during and after COVID-19 pandemic lockdown.

DETAILED DESCRIPTION:
Research describing training load management during COVID-19 enforced home training in professional tennis players is lacking. Therefore, the main objective of this case series is to describe in detail the training load management and progression of three professional tennis players before, during and after COVID-19 pandemic lockdown.

ELIGIBILITY:
Inclusion Criteria:

* tennis players training in argentina

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Tennis players training in argentina
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Training load | 12 months
  session RPE

CONTACTS AND LOCATIONS:
Overall Officials: Diego Mendez, PT, Principal Investigator — Kine Kinesiologia Deportiva y Funcional
Locations (1):
- KINÉ kinesiología deportiva y funcional, CABA, Argentina

IPD SHARING:
Plan to Share IPD: No